CLINICAL TRIAL: NCT06514053
Title: Discovering Prognostic Biomarkers for Pulpotomy Outcome in Permanent Mature Teeth With Irreversible Pulpitis
Brief Title: Prognostic Biomarkers for Pulpotomy Outcome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Zhang Chengfei, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW 23-133
Record Dates: First submitted 2024-04-17; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Pulpitis - Irreversible

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Full pulpotomy (Active Comparator)
  Interventions: Procedure: Full pulpotomy
- Root canal treatment (Active Comparator)
  Interventions: Procedure: Root canal treatment

INTERVENTIONS:
Procedure: Full pulpotomy — A full pulpotomy will be performed by removing the entire roof of the pulp chamber and the remaining pulp tissue will be covered by Biodentine.
  Arms: Full pulpotomy
Procedure: Root canal treatment — The regular procedure of root canal treatment will be performed on teeth with irreversible pulpitis
  Arms: Root canal treatment

SUMMARY:
This study will recruit 180 molars diagnosed with irreversible pulpitis. Full pulpotomy will be performed on 120 teeth, while RCT (root canal treatment) will be conducted on another cohort of 60 teeth as the control for assessing long-term outcomes. Additionally, 12 blood samples and pulp tissues from healthy teeth receiving elective RCT will be collected as the controls. The first pulpal blood sample will be collected after caries removal and pulp exposure. Subsequently, the entire coronal pulp tissue will be removed and collected for histological examination, image-based spatial and scRNA-seq analyses. A second pulpal blood sample will be collected from the radicular pulp tissue. Both blood samples will be used to profile the inflammation-related biomarkers through multiplex immunoassays. The remaining pulp tissue will be covered by Biodentine and restored with resin-based composite. Pulpotomy treatment outcomes will be evaluated clinically and radiographically at 6 and 12 months. The biomarkers identified in the pulpal blood and histology and the single-cell transcriptomes of the coronal pulp will be compared with the treatment "success" and "failure" groups upon one year. The outcome of RCT will be compared with that of full pulpotomy at 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Permanent molars showing clinical and radiographic evidence of a deep carious lesion (extend to the three-quarters thickness of dentine radiographically) extending close to the pulp chamber
* Clinical diagnosis of irreversible pulpitis, including spontaneous pain, lingering pain with cold stimulation, no or mild tenderness to percussion, normal apical tissue or widening of the periodontal ligament space but with no signs of periapical periodontitis (i.e., PAI score 1 or 2)
* Positive response to cold and electric pulp test.

Exclusion Criteria:

* Tooth with no response to the cold and electric tests, presence of apical radiolucency (greater than periodontal widening), signs of canal calcification and resorption, history of trauma, unrestorable or nonfunctional teeth, and evidence of perio-endo lesion
* Intraoperative bleeding time is more than 10 minutes or less than 10 μL pulpal blood can be obtained
* Patients with a compromised immune status (such as HIV or organ transplant) or with any history of taking analgesics/antibiotics in the past one week.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Success rate | 2 years
  Success rate of full pulpotomy and RCT in teeth with irreversible pulpitis
Biomarkers | 2 years
  Quantitative descriptive analysis of the expression of biomarkers commonly found in tissue inflammation using multiplex immunoassay (Millipore, USA). The kits include targets as follows: sCD40L;EGF;Eotaxin;FGF-2;Flt-3 ligand;Fractalkine;G-CSF;GM-CSF;GROα;IFNα2;IFNγ;IL-1α;IL-1β;IL-1ra;IL-2;IL-3;IL-4;IL-5;IL-6;IL-7;IL-8;IL-9;IL-10;IL-12 (p40);IL-12 (p70);IL-13;IL-15;IL-17A;IL-17E/IL-25;IL-17F;IL-18;IL-22;IL-27;IP-10;MCP-1;MCP-3;M-CSF;MDC (CCL22);MIG;MIP-1α;MIP-1β;PDGF-AA;PDGF-AB/BB;RANTES;TGFα;TNFα;TNFβ;VEGF-A; MMP-1, -2, -7, -9, -10.

SECONDARY OUTCOMES:
Correlation | 2 years
  Correlation of biomarkers' expression to the outcome of full pulpotomy in teeth with irreversible pulpitis to identify objective prognostic biomarkers for full pulpotomy; biomarkers to investigate are described in Outcome 2

CONTACTS AND LOCATIONS:
Overall Officials: Chengfei Zhang, Principal Investigator — The University of Hong Kong
Locations (1):
- Clinical Research Centre, Faculty of Dentistry, The University of Hong Kong, Hong Kong, Hong Kong